CLINICAL TRIAL: NCT00885378
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Trial to Evaluate the Efficacy and Safety of 2.5 mg Saxagliptin, Twice Daily, in Combination With Metformin IR in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin IR Alone
Brief Title: Efficacy and Safety Study of Saxagliptin + Metformin Immediate Release (IR) Versus Metformin IR Alone in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV181-080; EUDRACT #: 2009-010224-25
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2011-12-16 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin plus metformin IR (Active Comparator)
  Interventions: Drug: Saxagliptin plus metformin IR
- Placebo plus metformin IR (Placebo Comparator)
  Interventions: Drug: Placebo plus metformin IR

INTERVENTIONS:
Drug: Saxagliptin plus metformin IR — Tablets, Oral, 2.5 mg, Twice daily, 12 weeks
  Other Names: BMS-477118; Onglyza
  Arms: Saxagliptin plus metformin IR
Drug: Placebo plus metformin IR — Tablets, Oral, Placebo, Twice daily, 12 weeks
  Arms: Placebo plus metformin IR

SUMMARY:
The purpose of this study is to compare the reduction in hemoglobin A1C (A1C) for participants taking saxagliptin in combination with metformin immediate release (IR) versus metformin IR alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 18-78 years of age
* Taking stable twice daily (BID) dosing of metformin IR (at least 1500 mg) for at least 8 weeks
* A1C: 7-10%
* C-peptide: ≥ 0.8 ng/mL
* Body mass index (BMI): ≤45 kg/m^2

Exclusion Criteria:

* Women of childbearing potential unable or unwilling to use acceptable birth control
* Women who are pregnant or breastfeeding
* Fasting plasma glucose (FPG) >270 mg/dL
* Significant cardiovascular history
* Symptoms of poorly controlled diabetes
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Insulin therapy within one year of screening
* Cardiovascular even within the prior 6 months
* New York Heart Association Stage III/IV congestive heart failure and/or known left ventricular ejection fraction <=40%
* Significant history of renal or hepatic disease
* History of a psychiatric disorder, alcohol or drug abuse within the previous year
* Treatment with potent CYP3A4 inhibitors or inducers
* Immunocompromised participants
* Active liver disease or clinically significant abnormal hepatic, renal , endocrine, metabolic, or hematological screening tests

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (25):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Southland Clinical Research Center, Inc., Fountain Valley, California
  - Torrance Clinical Research, Lomita, California
  - Ritchken & First M.D.'S, San Diego, California
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Family Care Associates Of Nw Florida, Chipley, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Nextphase Clinical Trials, Inc., Miami, Florida
  - Middle Georgia Drug Study Center, Llc, Perry, Georgia
  - Louisiana Heart Center Research, Slidell, Louisiana
  - Jackson Clinic, Rolling Fork, Mississippi
  - Community Health Care Of Manchester, Akron, Ohio
  - Midwest Regional Research, Inc., Bellbrook, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - Newark Physician Associates, Newark, Ohio
  - Integris Family Care South, Oklahoma City, Oklahoma
  - Integris Family Care Yukon, Yukon, Oklahoma
  - Williamette Valley Clinical Studies, Eugene, Oregon
  - Integrated Medical Group Pc/Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Southeastern Research Associates, Inc, Taylors, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Village Family Practice, Houston, Texas
  - Southwest Clinical Research Centers, Llc, Pearland, Texas
  - Jolene K. Berg, Md., Dgd Research, Inc., San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
- Germany (7):
  - Local Institution, Ludwigshafen
  - Local Institution, Magdeberg
  - Local Institution, Pirna
  - Local Institution, Saarbrücken
  - Local Institution, Saarlouis
  - Local Institution, Tann
  - Local Institution, Wüstensachsen
- Hungary (5):
  - Local Institution, Balatonfüred, Hungary
  - Local Institution, Budapest
  - Local Institution, Eger
  - Local Institution, Szigetvár
  - Local Institution, Zalaegerszeg
- Puerto Rico (2):
  - Local Institution, Ponce
  - Local Institution, San Juan

REFERENCES:
- [Derived] White JL, Buchanan P, Li J, Frederich R. A randomized controlled trial of the efficacy and safety of twice-daily saxagliptin plus metformin combination therapy in patients with type 2 diabetes and inadequate glycemic control on metformin monotherapy. BMC Endocr Disord. 2014 Feb 24;14:17. doi: 10.1186/1472-6823-14-17. PMID 24565221
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at 43 sites in 4 countries (25 sites in the United States [US], 9 in Germany, 5 in Hungary, and 4 in Puerto Rico) received study medication and participated in this study.
Pre-assignment Details: Of the 166 subjects who entered the lead-in period, 6 discontinued: 3 withdrawal of consent, 1 poor/noncompliance, 1 adverse event (AE; abdominal pain secondary to partial small bowel obstruction), and 1 elevated liver enzymes that did not meet study exclusion criteria but was discontinued by the investigator.
Groups:
- Saxagliptin 2.5 mg + Metformin Immediate Release (IR): Saxagliptin 2.5 mg tablets orally (PO) plus a flexible metformin IR dose twice daily (BID).
- Placebo + Metformin IR: 2.5 mg placebo tablets PO BID plus flexible metformin IR dose.
Period: Overall Study
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Started | 74 (Number randomized.) | 86 (Number randomized.)
Completed | 66 | 78
Not Completed | 8 | 8
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Poor/Noncompliance | 2 | 2
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR | Total
Number analyzed (Participants) | 74 | 86 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.90 (10.35) | 56.60 (9.97) | 55.4 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 41 | 75
  Male | 40 | 45 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 64 | 80 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 56 | 105
  Hungary | 8 | 8 | 16
  Puerto Rico | 8 | 10 | 18
  Germany | 9 | 12 | 21
Mean Height [Mean (Standard Deviation); unit: cm] | 168.38 (9.56) | 167.77 (8.99) | 168.05 (9.23)
Mean Weight [Mean (Standard Deviation); unit: kg] | 95.85 (21.40) | 91.74 (19.87) | 93.64 (20.63)
Mean Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg / m^2] | 33.68 (5.94) | 32.51 (6.18) | 33.05 (6.08)
Participant Body Mass Index [Number; unit: Participants]
  < 30 kg / m^2 | 19 | 35 | 54
  >= 30 kg / m^2 | 55 | 51 | 106
Mean Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean time since the time of diagnosis of Type 2 Diabetes Mellitus.
  Years | 5.81 (6.37) | 6.17 (4.21) | 6.00 (5.30)
Mean Metformin Dose at Baseline [Mean (Standard Deviation); unit: mg] | 1911.5 (376.59) | 1855.8 (330.19) | 1881.6 (352.38)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Baseline and Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Mean change was adjusted for baseline.
Time Frame: Baseline, Week 12
Population: Randomized participants with a measurement at the specified timepoint with Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg / dL
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 73 | 84
mg / dL
  Mean Baseline | 164.22 (5.512) | 161.25 (4.624)
  Adjusted Mean Change from Baseline | -13.73 (4.51) | -4.22 (4.20)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin Immediate Release (IR) vs Placebo + Metformin IR; Test type: Superiority or Other; p = 0.1248, ANCOVA; ANCOVA model: post - pre = pretreatment; Mean Difference (Final Values) = -9.51, 95% CI 2-sided [-21.68 to 2.66], Standard Error of Mean 6.162 — Estimate = adjusted mean change for Saxagliptin - adjusted mean change for Placebo

2. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (A1C < 7.0%) at Week 12
Description: Adjusted for baseline. Calculated using the method by Zhang et al. (Zhang M, Tsiatis A, Davidian M. Improving efficiency of inference in randomized clinical trials using auxiliary covariates. Biometrics. Published online on January 11, 2008; Digital Object Identifier: 10.1111/j.1541-0420.2007.00976.x.)
Time Frame: Week 12
Population: Randomized participants with measurement at timepoint with LOCF.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 73 | 84
Percentage of Participants | 37.5 [27.4 to 47.6] | 24.2 [15.8 to 32.7]
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin Immediate Release (IR) vs Placebo + Metformin IR; Test type: Superiority or Other; Mean Difference (Final Values) = 13.2, 95% CI 2-sided [1.1 to 25.4] — Adjusted for baseline

3. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (A1C <= 6.5%) at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: Randomized participants with measurement at timepoint with LOCF.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 84
Percentage of Participants | 24.6 [15.1 to 34.1] | 10.7 [4.6 to 16.9]
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin Immediate Release (IR) vs Placebo + Metformin IR; Test type: Superiority or Other; Mean Difference (Final Values) = 13.8, 95% CI 2-sided [3.0 to 24.7] — Adjusted for baseline

4. Other Pre Specified Outcome: Participant Adverse Event (AE), Related AE, Serious Adverse Event (SAE), Related SAE, and Discontinued Due to AEs Summary
Description: AE = any new untoward medical occurrence/worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment.SAE = any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Treatment-related=Possible, Probable, or Certain relationship to drug.
Time Frame: Week 1 to Week 12; AEs are included up to the last treatment day + 1 day or the last visit in the double-blind (DB) period. SAEs are included up to the last of 1) the last treatment day + 30 days or 2) the last visit day + 30 days in the DB period.
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
Participants
  At Least 1 AE | 19 | 34
  At Least 1 Related AE | 1 | 3
  Deaths | 0 | 0
  At Least 1 SAE | 1 | 1
  At Least 1 Related SAE | 0 | 0
  Discontinued Due to SAEs | 0 | 0
  Discontinued Due to AEs | 0 | 0

5. Other Pre Specified Outcome: Participants With Reported Hypoglycemia AEs During Double-Blind Treatment Period
Description: Hypoglycemic Events are based upon the Saxagliptin Predefined List of Events, which included hypoglycemia, blood glucose decreased, and hypoglycemic unconsciousness.
Time Frame: Week 1 to Week 12; AEs are included up to the last treatment day + 1 day or the last visit in the DB period. SAEs are included up to the last of 1) the last treatment day + 30 days or 2) the last visit day + 30 days in the DB period.
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
Participants | 4 | 1

6. Other Pre Specified Outcome: Participants With Confirmed Hypoglycemia
Description: Confirmed hypoglycemia was defined by a fingerstick glucose value <= 50 mg/dL with associated hypoglycemia symptoms.
Time Frame: as for outcome 5
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
Participants | 0 | 1

7. Other Pre Specified Outcome: Participant Electrocardiogram (ECG) Status at Baseline and Week 12
Description: Abnormal ECGs were defined as those not within the normal limits for the participant, according to the investigator. 'Shifted Normal to Abnormal' and 'Shifted Abnormal to Normal' references a change from measurements at Baseline to those at Week 12.
Time Frame: Baseline, Week 12
Population: All treated participants, excluding those with missing values.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 71 | 78
Participants
  Baseline Normal | 36 | 42
  Baseline Abnormal | 35 | 36
  Week 12 Normal | 39 | 50
  Week 12 Abnormal | 32 | 28
  Shifted Normal to Abnormal | 5 | 4
  Shifted Abnormal to Normal | 8 | 12

8. Other Pre Specified Outcome: Baseline and Mean Change From Baseline in Participant Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Baseline values reference the measurement for the cohort of participants evaluated at the given time point.
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: All treated participants. n= number of participants with measurement at time point.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
mm Hg
  Baseline SBP for Week 4 cohort (n=74, 84) | 128.89 (1.67) | 127.57 (1.53)
  Baseline DBP for Week 4 cohort (n=74, 84) | 78.99 (1.07) | 77.07 (1.05)
  SBP Change From Baseline at Week 4 (n=74, 84) | -0.47 (1.43) | 0.17 (1.16)
  DBP Change From Baseline at Week 4 (n=74, 84) | -0.81 (0.84) | 0.95 (0.86)
  Baseline SBP for Week 8 cohort (n=70, 81) | 128.33 (1.67) | 127.60 (1.57)
  Baseline DBP for Week 8 cohort (n=70, 81) | 78.87 (1.08) | 77.32 (1.03)
  SBP Change From Baseline at Week 8 (n=70, 81) | 0.60 (1.66) | -0.43 (1.48)
  DBP Change From Baseline at Week 8 (n=70, 81) | 0.37 (0.94) | 0.86 (0.93)
  Baseline SBP for Week 12 cohort (n=66, 77) | 128.18 (1.76) | 127.38 (1.56)
  Baseline DBP for Week 12 cohort (n=66, 77) | 78.85 (1.13) | 77.23 (1.06)
  SBP Change From Baseline at Week 12 (n=66, 77) | 1.59 (1.51) | 0.83 (1.26)
  DBP Change From Baseline at Week 12 (n=66, 77) | 1.03 (0.75) | 1.29 (0.85)

9. Other Pre Specified Outcome: Baseline and Mean Change From Baseline in Participant Heart Rate (HR)
Description: Baseline values reference the measurement for the cohort of participants evaluated at the given time point.
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: All treated participants. n= number of participants with measurement at time point.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
mm Hg
  Baseline HR for Week 4 cohort (n=74, 84) | 73.45 (1.072) | 73.77 (0.968)
  HR Change From Baseline at Week 4 (n=74, 84) | 0.97 (0.881) | 1.18 (0.778)
  Baseline HR for Week 8 cohort (n=70, 81) | 73.51 (1.091) | 73.56 (0.990)
  HR Change From Baseline at Week 8 (n=70, 81) | 2.70 (0.914) | 0.28 (0.727)
  Baseline HR for Week 12 cohort (n=66, 77) | 73.71 (1.142) | 73.55 (1.035)
  HR Change From Baseline at Week 12 (n=66, 77) | 0.61 (1.061) | 0.60 (0.866)

10. Primary Outcome: Mean Hemoglobin A1C (A1c) and Change From Baseline to Week 12
Description: Mean change was adjusted for baseline.
Time Frame: Baseline, Week 12
Population: Randomized participants with both a baseline value and post-baseline value (up to Week 12).
Measure: Mean (Standard Error); unit: Percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 84
Percentage of glycosylated hemoglobins
  Baseline | 7.92 (0.11) | 7.97 (0.09)
  Adjusted Mean Change From Baseline | -0.56 (0.09) | -0.22 (0.08)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg + Metformin Immediate Release (IR) vs Placebo + Metformin IR; Test type: Superiority or Other; p = 0.0063, ANCOVA — Between-group comparisons significant at alpha = 0.05, significance testing based on hierarchical testing; Adjusted mean difference for saxagliptin groups vs placebo at Week 12(LOCF) was adjusted for baseline; Standard Error of the Mean = -0.34, 95% CI 2-sided [-0.58 to -0.10] — difference between week t value - baseline value = baseline value + treatment

11. Other Pre Specified Outcome: Participants Experiencing Changes From Baseline in Laboratory Parameters That Met the Marked Abnormality Criteria
Description: A laboratory value was considered a marked abnormality if it is outside the pre-defined criteria for marked abnormality and the on-treatment value was more extreme (farther from the limit) than the baseline value. ULN=upper limit of normal; LLN=lower limit of normal.
Time Frame: Baseline, Week 12
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
Participants
  Hemoglobin < 8 g/dL | 0 | 0
  Hematocrit < 0.75 prior to dosing | 0 | 0
  Platelets < 50 x 10^9 c/L | 0 | 0
  Platelets > 1.5 x ULN | 0 | 0
  Leukocytes < 2 x 10^3 c/uL | 0 | 0
  Neutrophils < 1 x 10^3 c/uL | 1 | 0
  Eosinophils > 0.9 x 10^3 c/uL | 0 | 2
  Lymphocytes <= 0.75 x 10^3 c/uL | 1 | 0
  Alkaline Phosphatase >3x prior to dosing and > ULN | 0 | 0
  Aspartate Aminotransferase > 3x ULN | 1 | 0
  Aspartate Aminotransferase > 5x ULN | 0 | 0
  Alanine Aminotransferase > 3x ULN | 1 | 0
  Alanine Aminotransferase > 5x ULN | 0 | 0
  Total Bilirubin > 2 mg/dL | 0 | 0
  Total Bilirubin > 1.5x ULN | 0 | 1
  Blood Urea Nitrogen > 2x prior to dosing and > ULN | 0 | 0
  Creatinine > 2.5 mg/dL | 0 | 0
  Serum Sodium <0.9x pre-Rx and <= 130 mEq/ | 0 | 0
  Serum Sodium >1.1x pre-Rx and >= 150 mEq/L | 0 | 0
  Serum Potassium <=0.8x pre-Rx and <= 3.2 mEq/L | 0 | 0
  Serum Potassium >=1.2x pre-Rx and >= 6.0 mEq/L | 1 | 0
  Serum Chloride <90 mEq/L | 0 | 0
  Serum Chloride > 120 mEq/L | 0 | 0
  Albumin <0.9x LLN, or if pre-Rx<LLN use <0.75x | 0 | 0
  Creatinine Kinase > 5x ULN | 0 | 1
  Fasting Plasma Glucose < 50 mg/dL | 1 | 0
  Fasting Plasma Glucose > 500 mg/dL | 0 | 0
  Plasma Glucose Unspecified < 50 mg/dL | 0 | 0
  Plasma Glucose Unspecified > 500 mg/dL | 0 | 0

12. Other Pre Specified Outcome: Participants Experiencing Changes From Baseline in Urinalysis Parameters That Met the Marked Abnormality Criteria
Description: Marked abnormality criteria were urine protein: if pre-Rx=o use >=2, if pre-Rx =0.5 or 1 use >=3, if pre-Rx =2, use >=4; urine blood: if pre-Rx=0, use >=2, if pre-Rx=0.5 or 1, use >=3, if pre-Rx=2, use >=4; Urine red blood cell count (RBC): if pre-Rx=o use >=2, if pre-Rx =0.5 or 1 use >=3, if pre-Rx =2, use >=4; urine white blood cell count (WBC): if pre-Rx=o use >=2, if pre-Rx =0.5 or 1 use >=3, if pre-Rx =2, use >=4.
Time Frame: Baseline, Week 12
Population: All treated participants. N = number of participants analyzed and n = the number of participants with values available for each specific measurement.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) | Placebo + Metformin IR
Number analyzed (Participants) | 74 | 86
Participants
  Urine Protein (n=74, 84) | 0 | 0
  Urine Blood (n=74, 84) | 1 | 1
  Urine Red Blood Cells (n=7, 10) | 0 | 0
  Urine White Blood Cells (n=16, 18) | 2 | 2

ADVERSE EVENTS:
Arm/Group | Placebo + Metformin IR | Saxagliptin 2.5 mg + Metformin Immediate Release (IR)
Serious Adverse Events (participants affected / at risk) | 1/86 | 1/74
Other Adverse Events (participants affected / at risk) | 0/86 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin IR (N=86) | Saxagliptin 2.5 mg + Metformin Immediate Release (IR) (N=74)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤ 60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.